CLINICAL TRIAL: NCT05868720
Title: EFFECT OF RISPERIDONE vs ARIPIPRAZOLE ON OXIDATIVE STRESS IN PATIENTS WITH AUTISM SPECTRUM DISORDER: A RANDOMIZED CONTROLLED TRIAL
Acronym: versus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Debadatta Mohapatra, Assistant Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC/PG Thesis/2022-23/126
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: The Goal of This Trial is to to Compare the Effect of Risperidone vs Aripiprazole in Terms of Change in Serum Glutathione Level
MeSH Terms: interventions — Risperidone; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risperidone group (Experimental)
  Interventions: Drug: Risperidone, Aripiprazole
- Aripiprazole group (Experimental)
  Interventions: Drug: Risperidone, Aripiprazole

INTERVENTIONS:
Drug: Risperidone, Aripiprazole — The patients who are randomized to Risperidone group will receive Risperidone at a dose of 1mg/day during the study period that is for 6 weeks. The patients who are randomized to Aripiprazole group will receive Aripiprazole at a dose of 2mg/day during the study period that is for 6 weeks.

SUMMARY:
The goal of this Randomized Controlled Trial is to to compare the effect of Risperidone vs Aripiprazole in terms of change in serum Glutathione level in patients with Autism Spectrum Disorder over a period of 6 weeks.

The main questions it aims to answer are:

1. (Primary Outcome) Change in serum Glutathione levels following 6 weeks of intervention in both the arms
2. (Secondary Outcomes) Change in serum superoxide dismutase (SOD) levels following 6 weeks of intervention.

Change in ISAA score following 6 weeks of intervention. Change in ABC-C score following 6 weeks of intervention. • Adverse events reported in both groups

Details of intervention- One arm of the study population to get Risperidone 1mg/day for a total duration of 6 weeks and another arm to get Aripiprazole 2mg/day for a total duration of 6 weeks. Baseline assessment of Serum Glutathione, Serum SOD, ISAA scale, ABC-C scale will be done and same will be assesssed at 6 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Patients diagnosed with Autism Spectrum Disorder (according to ICD-11 DCR) under the age group of 18 years.
  * Legally authorized representative (LAR) giving voluntary written consent for participation in the study.

Exclusion Criteria:

* History of ADHD

  * History of any major genetic disorder/ storage disorder/ any special syndromes.
  * History of seizure disorder or any major medical or surgical disorders
  * Legally authorized representative (LAR) not giving voluntary written consent for participation in the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-05-02 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Change in serum Glutathione levels following 6 weeks of intervention in both the arms | 6 weeks
  Change in serum Glutathione levels following 6 weeks of intervention in both the arms

SECONDARY OUTCOMES:
Change in serum superoxide dismutase (SOD) levels following 6 weeks of intervention. | 6 weeks
Change in ISAA score following 6 weeks of intervention. | 6 weeks
Change in ABC-C score following 6 weeks of intervention. • | 6 weeks
Adverse events reported in both groups | 6 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hodges H, Fealko C, Soares N. Autism spectrum disorder: definition, epidemiology, causes, and clinical evaluation. Transl Pediatr. 2020 Feb;9(Suppl 1):S55-S65. doi: 10.21037/tp.2019.09.09. PMID 32206584
- [Result] Salari N, Rasoulpoor S, Rasoulpoor S, Shohaimi S, Jafarpour S, Abdoli N, Khaledi-Paveh B, Mohammadi M. The global prevalence of autism spectrum disorder: a comprehensive systematic review and meta-analysis. Ital J Pediatr. 2022 Jul 8;48(1):112. doi: 10.1186/s13052-022-01310-w. PMID 35804408
- [Result] Minshew NJ, Williams DL. The new neurobiology of autism: cortex, connectivity, and neuronal organization. Arch Neurol. 2007 Jul;64(7):945-50. doi: 10.1001/archneur.64.7.945. PMID 17620483
- [Result] Pandya CD, Howell KR, Pillai A. Antioxidants as potential therapeutics for neuropsychiatric disorders. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Oct 1;46:214-23. doi: 10.1016/j.pnpbp.2012.10.017. Epub 2012 Nov 2. PMID 23123357
- [Result] Salim S. Oxidative stress and psychological disorders. Curr Neuropharmacol. 2014 Mar;12(2):140-7. doi: 10.2174/1570159X11666131120230309. PMID 24669208